CLINICAL TRIAL: NCT02913352
Title: Randomized Trial for the Treatment of Recurrent Anterior Dislocation of the Shoulder: Latarjet Versus Modified Eden-Hybinette
Brief Title: Latarjet Versus Modified Eden-Hybinette for Anterior Shoulder Dislocation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Faculdade de Medicina de Jundiaí (Other)
Responsible Party: Principal Investigator, Mauro Gracitelli, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Latarjet vs Eden
Record Dates: First submitted 2016-09-16; First posted 2016-09-23 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Latarjet procedure (Active Comparator): Open Latarjet-Patte procedure. Surgery. Anterior glenoid bone graft from coracoid. Fixation with 2 screws.
  Interventions: Procedure: Latarjet procedure
- Modified Eden-Hybinette Procedure (Experimental): Surgery. Modified Eden-Hybinette surgery, with capsular repair on the iliac bone Anterior glenoid bone graft from iliac bone. Fixation with 2 screws.
  Interventions: Procedure: Modified Eden-Hybinette

INTERVENTIONS:
Procedure: Latarjet procedure — Open anterior glenoid bone graft from coracoid process
  Arms: Latarjet procedure
Procedure: Modified Eden-Hybinette — Open anterior glenoid bone graft from iliac bone crest, with capsular suture and screw fixation
  Arms: Modified Eden-Hybinette Procedure

SUMMARY:
Randomized clinical trial, parallel 1:1, comparing Latarjet to Modified Eden-Hybinette (iliac bone crest + capsular repair) for recurrent traumatic anterior glenohumeral dislocation.

DETAILED DESCRIPTION:
The Latarjet technique has proven reliable for the treatment of dislocations, with lower recurrence rates (5%) even in the presence of bone lesions. This technique allows a stable fixation of the graft, with 2 screws, and the dynamic effect of the conjoint tendon, the sling effect. However, several complications are described, such as neurological injuries, nonunion and graft resorption. Hamel et al, showed that vascularization of the coracoid graft is impaired during the course of Latarjet procedure. Together with the small thickness of the coracoid, it may justify its high rate of resorption.

The Eden-Hybinette surgery does not have the potential advantages of the sling effect. However, it allows a better restoration of the area of the glenoid, without the risks related to the coracoid osteotomy. All clinical studies about the different bone grafting techniques have a low quality. Furthermore, there is no comparative study of the techniques of Latarjet and Eden-Hybinette.

ELIGIBILITY:
Inclusion Criteria:

* History of one or more previous episodes of traumatic glenohumeral dislocation;
* Anterior glenoid bone loss superior to 20% of its diameter, regardless of the ISIS score;
* Recurrence of glenohumeral dislocation in cases previously treated with arthroscopic Bankart repair, regardless of the ISIS score and severity of bone lesion of the glenoid;
* Borderline bipolar bone lesions:
* Instability Severity Index Score of (ISIS) greater than or equal to 4 points, with anterior glenoid bone loss (bone Bankart lesion) greater than 13.5% of their diameter, measured by the method described by Sugaya et al.;
* Hill-Sachs lesion and glenoid considered "off-track".

Exclusion Criteria:

* Hill-Sachs lesion greater than 40% of the humeral head diameter (measured by the preoperative CT);
* Untreated seizures;
* Previously diagnosed rotator cuff complete tear;
* Fractures of the proximal humerus (except for Hill-Sachs lesions);
* Multidirectional instability;
* Advanced glenohumeral osteoarthritis (grade 3 Samilson and Pietro)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09-01; Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability Index (WOSI) | 2 years
  Instability score

SECONDARY OUTCOMES:
ROWE score | 2 years
Visual analog scale (VAS) for shoulder pain | 2 years
VAS for iliac pain | 6 weeks
VAS for iliac pain | 3 months
VAS for iliac pain | 2 years
Single Assessment Numeric Evaluation (SANE) | 2 years
Dislocation recurrence rate | 2 years
Rate of complications and reoperations | 2 years
Kible scale for Scapular movement | 2 years
  Scale for scapular positioning. Clinical measurement
Categoric evaluation for scapular movement | 2 years
  Video evaluation for normal or dyskinesis of the scapula movement
Tomographic evaluation | 2 years
  Graft union, graft position and resorption
Radiographic evaluation | 2 years
  Graft union, graft position and resorption
Degree of Shoulder Involvement in Sports (DOSIS ) scale | 2 years
  return to sport scale

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Ortopedia e Traumatologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided